CLINICAL TRIAL: NCT02488863
Title: Neuroimaging Age-related Versus Pain-related Changes in Pain Modulation
Brief Title: NEPAL (Neuromodulatory Examination of Pain and Mobility Across the Lifespan)
Acronym: NEPAL
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201401056-N; K01AG048259 (NIH); P30AG059297 (NIH); Pepper Grant (Other Grant/Funding Number: National Institute of Health)
Record Dates: First submitted 2014-12-23; First posted 2015-07-02 (Estimated); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Musculoskeletal Pain; Pain, Chronic
Keywords: Older adults; Chronic Pain; Musculoskeletal
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Older Adults with Musculoskeletal Pain: Older adults (60+ years old) experiencing musculoskeletal pain will undergo: MRI Neuroimaging, Quantitative Sensory Testing, Physical and Cognitive Function Testing, and questionnaire batteries.
  Interventions: Other: MRI Neuroimaging; Other: Quantitative Sensory Testing; Other: Questionnaires; Other: Physical and Cognitive Function Testing
- Older Adults without Musculoskeletal Pain: Older adults (60+ years old) not experiencing musculoskeletal pain will undergo: MRI Neuroimaging, Quantitative Sensory Testing, Physical and Cognitive Function Testing, and questionnaire batteries.
  Interventions: Other: MRI Neuroimaging; Other: Quantitative Sensory Testing; Other: Questionnaires; Other: Physical and Cognitive Function Testing
- Young Controls: Healthy young adults (18-25 years old) not experiencing musculoskeletal pain will undergo: MRI Neuroimaging, Quantitative Sensory Testing, Physical and Cognitive Function Testing, and questionnaire batteries.
  Interventions: Other: MRI Neuroimaging; Other: Quantitative Sensory Testing; Other: Questionnaires; Other: Physical and Cognitive Function Testing

INTERVENTIONS:
Other: MRI Neuroimaging — MRI scans utilized to measure the structural and functional integrity of the brain.
  Other Names: Functional Magnetic Resonance Imaging (fMRI)
Other: Quantitative Sensory Testing — Vibratory Detection Thresholds; Tactile Detection Thresholds; Thermal Detection Thresholds, Pain Thresholds, and Temporal Summation; Allodynia and Temporal Summation; Punctate Pain Testing and Temporal Summation; and Pressure Pain Thresholds.
  Other Names: QST
Other: Questionnaires — The Modified Mini-Mental State Examination (3MS), the Montreal Cognitive Assessment (MoCA), the Center for Epidemiologic Studies Depression Scale (CES-D), the Geriatric Depression Scale (GDS), the Edinburg Handedness Inventory, the Ten-Item Personality Inventory (TIPI), the Pittsburgh Sleep Quality Index (PSQI), the state and trait versions of the State-Trait Anxiety Inventory (STAI), the state and trait versions of the Positive and Negative Affect Schedule (PANAS), pain questionnaires (the Graded Chronic Pain Scale (GCPS), the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Pain-Detect, the short-form McGill Pain Questionnaire (SF-MPQ-2), and the Coping Strategies Questionnaire-Revised (CSQ-R)), a standardized paper and pencil cognitive battery (Hopkins Verbal Learning Test (HVLT), Trail Making A&B, Boston Naming Test, Controlled Oral Word Association Test (COWAT), Stroop Interference Test, Ruff Figural Fluency Test, and Raven's Progressive Matrices Test).
Other: Physical and Cognitive Function Testing — Upper Limb Isometric Strength, Short Physical Performance Battery (SPPB), GAITRite Instrumented Walking, Galvanic Skin Response, Knee Extension Isokinetic Strength, the Pepper Assessment Tool for Disability (PAT-D), and an electronic NIH Toolbox Cognitive Battery.

SUMMARY:
Musculoskeletal pain represents the leading cause of disability worldwide. It has been traditionally attributed to peripheral mechanisms, but peripheral damage, inflammation, and psychological factors have failed to significantly account for the presence, absence, or severity of chronic musculoskeletal pain (CMP). Recent studies show that individuals with CMP exhibit dysfunctional pain modulation supporting a significant central nervous system (CNS) contribution. However, the CNS mechanisms underlying these changes in pain modulation are not currently known, nor is their relation to clinical pain progression. The proposed pilot examines brain circuits recently described in predicting the transition from acute to chronic pain, in predicting clinical and experimental pain changes as well as physical performance and mobility changes in older persons with musculoskeletal pain over a one year period. The findings will provide novel and important information regarding the mechanisms underlying aberrant pain processing and its functional consequences in older adults with musculoskeletal pain. The information learned can be subsequently used to target treatment and prevention strategies in future studies of older adults. The central hypothesis is that increased functional and structural connectivity of cortico-striatal regions will be significantly associated with baseline clinical and experimental pain and decreased physical function in persons with CMP and will account for more rapid clinical pain and disability progression over time.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain (CMP) is the most common, non-malignant disabling condition that affects at least one in four older people. The most common painful musculoskeletal conditions among older adults are osteoarthritis, low back pain, fibromyalgia, chronic shoulder pain, knee pain, myofascial pain syndrome and previous fracture sites. Recent studies demonstrate generalized alterations of pain processing among older individuals with CMP. An improved understanding of the mechanisms underlying CMP-related changes in pain modulation will provide a basis for the development of targeted preventive and rehabilitative strategies. In light of evidence emphasizing plasticity of white matter connections, and the potential pain relieving effects of non-invasive brain stimulation interventions, it seems reasonable to identify these connections as potential targets for future treatment approaches. Given the expected growth of the older population, such strategies could have a monumental impact in reducing healthcare expenditures and improving the quality of life of older adults.

ELIGIBILITY:
Inclusion Criteria:

* older adults over 60 years of age with and without musculoskeletal pain
* healthy young adults between the ages of 18-25

Exclusion Criteria:

* pregnant women
* history of alcohol/drug abuse in the past
* known intra-cerebral pathology or epilepsy
* significant cognitive impairment as evidenced by the 3MS
* hospitalizations for mental health reasons in the past year
* not meeting MRI screening requirements (implants, prosthesis, artificial limb/joint, shunt, metal rods, hearing aid, claustrophobia or anxiety)
* chronic/current use of narcotic medications
* serious systemic (uncontrolled diabetes; self reported A1C>7), neurological , or cardiovascular disease (uncontrolled hypertension >155/90)
* liver or kidney disease
* inability to consent for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults (60+ years old) who experience musculoskeletal pain as well as those who do not experience musculoskeletal pain; healthy young adults (18-25 years old).
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-07; Primary Completion 2024-02-04 (Actual); Study Completion 2024-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yenisel Cruz-Almeida, MSPH, PhD, Principal Investigator — University of Florida
Locations (4):
- United States (4):
  - UF & Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida
  - UF Health Science Center, Gainesville, Florida
  - Clinical Translational Research Building, Gainesville, Florida
  - McKnight Brain Institute of the University of Florida, Gainesville, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Older Adults With Musculoskeletal Pain | Older Adults Without Musculoskeletal Pain | Young Controls
Started | 53 | 22 | 30
Completed | 44 | 22 | 20
Not Completed | 9 | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Older Adults With Musculoskeletal Pain | Older Adults Without Musculoskeletal Pain | Young Controls | Total
Number analyzed (Participants) | 53 | 22 | 30 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 30 | 30
  >=65 years | 53 | 22 | 0 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 10 | 16 | 61
  Male | 18 | 12 | 14 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African American | 5 | 0 | 1 | 6
  Race/Ethnicity: Asian | 0 | 0 | 3 | 3
  Race/Ethnicity: Caucasian | 46 | 22 | 17 | 85
  Race/Ethnicity: Hispanic | 1 | 0 | 7 | 8
  Race/Ethnicity: Pacific Islander | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 53 | 22 | 30 | 105

OUTCOME MEASURES:

1. Primary Outcome: Short Physical Performance Battery (SPPB)
Description: The Short Physical Performance Battery (SPPB) Total Score is a measure of physical function. It is calculated by summing three measures of lower-extremity function: standing balance (side-by-side, semi-tandem, and tandem stance), 4-meter walking speed, and ability to rise from a chair. Each task is rated on a 0-4 scale, with increasing scores indicating better physical performance. The SPPB Total scores range from 0-12.
Time Frame: At baseline-physical function visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older Adults With Musculoskeletal Pain | Older Adults Without Musculoskeletal Pain | Young Controls
Number analyzed (Participants) | 44 | 22 | 20
score on a scale | 10.95 (1.10) | 10.82 (1.87) | 11.75 (0.64)
Statistical Analysis 1: Comparison: Older Adults With Musculoskeletal Pain vs Older Adults Without Musculoskeletal Pain vs Young Controls; H0: mean(SPPB_older_pain) = mean(SPPB_older_no pain) = mean(SPPB_younger); Test type: Other — ANOVA; p = 0.0561, ANOVA

ADVERSE EVENTS:
Time Frame: Each participant was assessed over their time in the study, about 2 weeks
Arm/Group | Older Adults With Musculoskeletal Pain | Older Adults Without Musculoskeletal Pain | Young Controls
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/22 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/22 | 0/30
Other Adverse Events (participants affected / at risk) | 2/53 | 0/22 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Older Adults With Musculoskeletal Pain (N=53) | Older Adults Without Musculoskeletal Pain (N=22) | Young Controls (N=30)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Participant reported a red mark left from the thermal stimulation during the MRI visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT02488863/Prot_001.pdf
  • Informed Consent Form (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT02488863/ICF_000.pdf